CLINICAL TRIAL: NCT05116072
Title: Efficacy and Safety of Total Pancreatectomy With Intraportal Islet Autotransplantation for Resectable Adenocarcinoma of the Cephalic Region of the Pancreas at High-risk of Postoperative Fistula and Requiring Systemic Adjuvant Chemotherapy
Brief Title: Efficacy and Safety of TPIAT for Resectable Adenocarcinoma of the Pancreas Region at High Risk of Postoperative Fistula
Acronym: TPIAT-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019_27; 2021-A00136-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-10-11; First posted 2021-11-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma of the Pancreas; Adenocarcinoma of the Duodenum; Ampullary Adenocarcinoma
Keywords: the cephalic region of the pancreas; total pancreatectomy; postoperative pancreatic fistula; islet transplantation; adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients benefited from total pancreatectomy for resectable adenocarcinoma of the cephalic region at high risk of postoperative pancreatic fistula, with intaportal/intramuscular islet autotransplantation
  Interventions: Procedure: total pancreatectomy; Biological: intraportal islet autotransplantation

INTERVENTIONS:
Procedure: total pancreatectomy — The total pancreatectomy will be performed in two steps: The pancreatectomy will begin by a standard pancreaticoduodenectomy procedure.
  The section margin will be sent for intraoperative histological analysis to confirm the absence of invasion of the left remnant pancreas.
  When absence of tumor invasion is confirmed and the high-risk of postoperative pancreatic fistula is validated intraoperatively, the extended left distal pancreatectomy will be performed, with splenic preservation when possible.
  Then, the left side of the pancreas will be resected and cooled (4-6°) in the preservation solution and shipped to Lille Biotherapy platform to perform islet isolation and purification. The reconstruction after total pancreatectomy will be done as usually performed by center expert surgeon.
Biological: intraportal islet autotransplantation — The final islet preparation will be cultured and shipped 48 hours after total pancreatectomy from the Lille laboratory to the surgical center, and finally transplanted into the patient through a venous catheter placed in the portal trunk (91% of the total islet mass) and at the same time, a small fraction of the isolated islet (5% of the total islet mass) will be transplanted into the forearm muscle.

SUMMARY:
Curative management of locally resectable invasive adenocarcinomas located in the cephalic region of the pancreas (pancreas, duodenum and ampulla of Vater) requires a pancreaticoduodenectomy followed by adjuvant chemotherapy. Pancreaticoduodenectomy is a major surgery that often leads to major complications including approximately 20% of relevant clinical postoperative pancreatic fistula.

Postoperative complications following pancreaticoduodenectomy can lead to early discontinuation of the complete oncologic strategy, i.e., chemotherapy for malignancy is performed in only about a third of patients who experienced a grade C fistula.

A total pancreatectomy rather than a pancreaticoduodenectomy is an alternative procedure that involves the complete and definitive resection of all pancreatic tissue, eliminating any risk of postoperative pancreatic fistula but is associated with unavoidable endocrine insufficiency and potentially severe metabolic complications, such as "brittle diabetes".

Total Pancreatectomy following by intraportal Islet AutoTransplantation (TPIAT) can prevent "brittle diabetes" and improve the quality of life. The endocrine islets can be isolated from the pancreatic surgical specimen with standardized procedures and transplanted in the liver through intraportal infusion, in absence of immunosuppression and allow adequate control of glucose metabolism with a reduced need for exogenous insulin and an effective graft function in 70% of cases at 3 years Thereby, the investigators hypothesize that total pancreatectomy with intraportal Islet autotransplantation rather than classical pancreaticuduodenectomy, in patients with high-risk of postoperative fistula will increase the rate of complete access to adjuvant chemotherapy, while maintaining an adequate metabolic control.

DETAILED DESCRIPTION:
Curative management of locally resectable invasive adenocarcinomas located in the cephalic region of the pancreas (pancreas, duodenum and ampulla of Vater) requires a pancreaticoduodenectomy followed by adjuvant chemotherapy. Pancreaticoduodenectomy is a major surgery that often leads to major complications including approximately 20% of relevant clinical postoperative pancreatic fistula. Severe postoperative pancreatic fistulas (grade C) require reoperation or lead to organ failure and/or mortality. In an extensive international registry study of pancreaticoduodenectomy procedures, chemotherapy for malignancy was performed in only about 33% (on time in 7% and delayed in 25.6 % of patients) and never delivered in about 67,4 % of patients who experienced a grade C fistula. Therefore, postoperative complications following pancreaticoduodenectomy can lead to early discontinuation of the complete oncologic strategy.

A total pancreatectomy rather than a pancreaticoduodenectomy is an alternative procedure that involves the complete and definitive resection of all pancreatic tissue, eliminating any risk of postoperative pancreatic fistula.

Total pancreatectomy could represent a major shift in the surgical management of patients with a high-risk of postoperative fistula by eliminating the life-threatening risk associated with fistula and by increasing the opportunity to initiate and to complete adjuvant chemotherapy without delay.

However, total pancreatectomy is associated with unavoidable endocrine insufficiency and potentially severe metabolic complications, such as "brittle diabetes".

Total Pancreatectomy with intraportal Islet AutoTransplantation (TPIAT) is currently performed in patients with chronic pancreatitis under chronic pain failing endoscopic treatment and dependent on long-term opioid treatment.

Therefore, islet autotransplantation following total pancreatectomy can prevent "brittle diabetes" and improve the quality of life.

The endocrine islets can be isolated from the pancreatic surgical specimen with standardized procedures and transplanted in the liver through intraportal infusion, in absence of immunosuppression and allow adequate control of glucose metabolism with a reduced need for exogenous insulin and an effective graft function in 70% of cases at 3 years

Thereby, the investigators hypothesize that total pancreatectomy with intraportal Islet autotransplantation rather than classical pancreaticuduodenectomy, in patients with high-risk of postoperative fistula will increase the rate of complete access to adjuvant chemotherapy, while maintaining an adequate metabolic control.

ELIGIBILITY:
Inclusion criteria

Inclusion criteria are composed of preoperative conditions validated by intraoperative confirmation to plan an exit of the protocol if the pancreas does not finally appear with a high-risk of CR-POPF.

* Age ≥ 18 years
* Locale resectable invasive adenocarcinomas located in the cephalic region of the pancreas documented by endoscopic ultrasonography with fine-needle aspiration biopsy
* pancreatic adenocarcinoma;
* duodenal adenocarcinoma;
* ampullary adenocarcinoma;
* and IPMNs with adenocarcinoma degeneration;
* A potentially curative strategy with primary tumor resection approved by a multidisciplinary expert team
* A high-risk of CR-POPF

  1. Suspected during preoperative evaluation by the presence of 2 or more of the following criteria (screening criteria of inclusion) : sex male;an obesity (BMI ≥ 30 kg/m2);a main pancreatic duct diameter ≤ 3 mm on preoperative endoscopic ultrasonography a visceral obesity (i.e. a visceral fat area > 84 cm2) ; a sarcopenia (i.e. a skeletal muscle index < 43 cm2/m2 in men with a BMI of <25 kg/m2 or <53 cm2/m2 in men with a BMI of ≥25 kg2/m2, and <41 cm2/m2 in women)
  2. and validated during intraoperative evaluation (finale inclusion) by a probability score above or equal to 20% on the validated updated alternative Fistula Risk Score ua-FRS for pancreaticoduodenectomy (ua-FRS) based of pancreas texture, duct size, BMI, sex .
* Women of childbearing potential should only be included after a confirmed menstrual period, and a negative highly sensitive urine or serum pregnancy test and must agree to be subjected to a monthly pregnancy test (urine or blood) until the end of the relevant systemic exposure to chemotherapy agents, in accordance with current CTFG recommendations (Recommendations related to contraception and pregnancy testing in clinical trials);
* Women of child-bearing potential and male subjects must agree to use a birth control methods which may be considered as highly effective (failure rate of less than 1% per year ) as recommended by the CTFG (Cinical Trials Facilitation and Coordination Group, version 1.1). These recommandations related to contraception and pregnancy testing in clinical trials suggested such method (see below) that will be use during chemotherapy exposure for included women of child-bearing potential and woman of child-bearing potential when partner of included male : combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal) ; progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable) ; intrauterine device (IUD) ; intrauterine hormone-releasing system ( IUS) ; bilateral tubal occlusion; vasectomised partner ;sexual abstinence For included male partner of a women of child-bearing potential, contraception with condom.

Contraception will be perform during the relevant systemic exposure to chemotherapy agents and will be extended by 6 months for women of childbearing potential and by 1 month for men included as recommended by the CTFG

* Patient covered by a health insurance system
* Patient who provides a written informed consent to participate to the study

Exclusion criteria

* Patient will be screened and excluded if they present a preoperative diabetes defined by a stimulated C-peptide < 0.5 ng/mL relative to blood glucose > 2 g/dL, at 2 hours in post prandial
* Patients with a known or highly suspected genetic syndrome associated with a risk of pancreatic adenocarcinoma: familial pancreatic cancer, multiple familial melanoma, Peutz-Jeghers syndrome, hereditary chronic pancreatitis, cystic fibrosis, familial breast Ovarian Cancer, Lynch syndrome, adenomatous polyposis family, Li Fraumeni syndrome, Multi-endocrine disorder type I;
* Multifocal pancreatic adenocarcinomas identified during preoperative evaluation;
* Performance status and comorbidity profile inappropriate for a major abdominal surgery;
* Contraindication for autologous islet intraportal transplantation
* Current or indicated/scheduled neoadjuvant chemotherapy;
* Extra pancreatic metastasis identified during preoperative evaluation (high-definition cross-sectional imaging with thorax-abdomen-pelvis multi-detection computed tomography or abdominal MRI with T1, T2 and diffusion weighted sequences) or during intraoperative assessment (clinical examination and ultrasonography);
* Need for complex vascular reconstructions (endovascular treatment or release of the arcuate ligament will be not considered as complex vascular reconstructions), major vein reconstructions will exclude the patients because of the over-risk of portal thrombosis following islet intraportal infusion.
* evident macroscopically or biologically proved post biliary drainage pancreatitis that jeopardize islet isolation
* Known infection or positive serology performed at screening for human immunodeficiency virus (HIV) infection, Hepatitis B or C virus infection, HTLV infection or syphilis infection.
* Active infection for SARS-CoV-2 virus (positive PCR), which will require rescheduling of the intervention 30 days later.
* Pregnant or breastfeeding woman
* Dihydropyrimidine dehydrogenase total deficiency
* Ethics / regulatory criteria :

  * Person unable to understand purposes, benefits and risks of the study and/or unable to provide a written informed consent.
  * Person unable to comply with the whole study schedule.
  * Person not covered by a health insurance system.
  * Person kept in detention and/or receiving psychiatric medical care and/or patients admitted in a social or medical sanatorium.
  * Person in an emergency situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
the rate of patients who have completed the chemotherapy planned | at postoperative month 12 following surgery.
  success is defined when patients treated with TPIAT will have completed the adjuvant systemic chemotherapy initially approved and planned by the local multidisciplinary expert team according to current international guidelines

SECONDARY OUTCOMES:
Rate of postoperative complications related to total pancreatectomy. | At 3 months following surgery.
  postoperative complication will be evaluated with Dindo Clavien classification
Rate of complications related to islet transplantation during the study | through study completion, at 36 months following surgery.
  complications related to islet transplantation will be reported according to CTCAE v5.0.
Mean time (in weeks) between TPIAT and adjuvant systemic chemotherapy. | through study completion, at 36 months following surgery.
  the time in weeks between TPIAT procedure and the adjuvant systemic chemotherapy will be reported
Rate of patients with cancer recurrence | at 3, 6, 9, 12, 24, and 36 months following surgery.
  The cancer recurrence will be assessed according standard of care imaging (Thorax multi-detection Computed Tomography, Abdomino-pelvis imaging : Mutli-detection Computed Tomography OR Magnetic Resonance Imaging) through the follow up using the Recist 1.1 criteria
Postoperative diabetes and pancreatic endocrine insufficiency following pancreatic surgery as recommended by the best standard care will be evaluated | functions before surgery and at day 7 and at 3, 12, 24 and 36 months following surgery.
  Postopeartive diabetes and exocrine insufficiency will be evaluated with clinical examination (symptoms, Pancreatic enzyme replacement therapy dosage, Diabetes medication : non insulin medication, insulin (daily insuline dosage UI/kg); blood samples (Fasting C-peptide and glycemia, Post-prandial C-peptide and glycemia, HbA1C (%))
EORTC QLQ-C30 core with it specific pancreatic module QLQ -PAN26 | at 3, 12, 24 and 36 months following surgery.
  EORTC QLQ-C30 and QLQ -PAN26 are self-completion questionnaires specific to cancer patients quality of life and pancreatic cancer patients quality of life
Rate of adverse events | through study completion, at 36 months following surgery.
  adverse events will be reported according to CTCAE v5.0 and classified according to their suspected or confirmed reason (i.e. chemotherapy, intraportal islet transplantation, pancreatic surgery)
Mortality rate | at day 7 and at 3, 12, 24 and 36 months following surgery.
  patient's death will be reported
islet transplantation success rate defined by CIT criteria | at 3, 12, 24 and 36 months following surgery.
  Islet transplantation succes status is defined by HbA1C < 7% AND no severe hypoglycemic event
islet transplantation success rate defined by IGLS 2.0 criteria | at 3, 12, 24 and 36 months following surgery.
  Islet transplantation succes status is defined by HbA1C < 7% AND no severe hypoglycemic event AND C-peptide ≥ 0.2 ng/mL
Primary islet Graft Function | at 1 month following TPIAT.
  Defined by the Beta 2 score calculated at 1 month post TPIAT using blood sample with fasting C peptide and glycemic, HbA1c and exogenous insuline requirement
mean number of Serious Hypoglycemic Event (SHE) since last visit | at day 7 and months 3, 12, 24 and 36 following surgery.
  Serious Hypoglycemic Event is defined as one requiring third-party assistance or resulting in hospitalization in an intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: François PATTOU, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France